CLINICAL TRIAL: NCT01917526
Title: The Performance Comparison of Two Oxygen Delivery Devices [Nasal Cannula and Mask] Used After General Anesthesia.
Brief Title: The Performance of Two Oxygen Delivery Devices Used After General Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 066/2556 (EC3)
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Hypoxemia
Keywords: Oxygen; PACU; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen mask (Active Comparator): Oxygen mask with oxygen flow 5 L/min will be given to allocated post general anesthesia patients. The incidence and causes of hypoxemia will be recorded.
  Interventions: Device: oxygen mask
- Oxygen cannula (Active Comparator): Oxygen cannula with oxygen flow 4 L/min will be given to allocated post general anesthesia patients. The incidence and causes of hypoxemia will be recorded.
  Interventions: Device: oxygen cannula

INTERVENTIONS:
Device: oxygen mask
  Other Names: Oxygen mask or simple mask
  Arms: oxygen mask
Device: oxygen cannula
  Arms: Oxygen cannula

SUMMARY:
After general anesthesia, there are the risks for airway obstruction, hypoventilation, atelectasis, ventilation-perfusion mismatch, hypercarbia and hypoxemia,so oxygen supplement in PACU seems necessary.

This study aim is to compare the two methods of oxygen supplement which are 1.nasal cannula at O2 flow 4 L/min. 2.oxygen mask with O2 flow 5 L/min. The hypothesis in this study is the 2 methods can equally provide effective oxygen supplement to prevent anesthesia-related hypoxemia. Choosing nasal cannula would be reasonable because it is cheaper and more comfortable to patient.

DETAILED DESCRIPTION:
The incidence and causes of hypoxemia in PACU will be identified, if necessary, a higher flow or changing oxygen delivery system can be used to prevent and treat hypoxemia. If any patients fail from oxygen weaning protocol in PACU and need longer oxygen therapy at ward, the duration of oxygen therapy will be recorded and also the compliance with oxygen delivery devices.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Age 18-70 years
* American Society of Anesthesiology (ASA)physical status 1-3
* Elective case

Exclusion Criteria:

* ASA physical status class 4 or more
* Unstable pulmonary diseases
* BMI > 35 kg/m2
* oxygen saturation < 94% when breathing in room air
* Respiratory muscle weakness eg.myasthenia gravis
* Central nervous system abnormalities eg.drowsiness, hypoventilation
* Patients who have been intubated or needed ventilatory support before operation
* Plan to remain intubated after the operation
* Intracranial, intrathoracic and upper abdomen surgery
* Patients who nasogastric tube is inserted
* Airway problems eg. sinusitis
* Nasal cavity related surgery or nasal packing eg. endoscopic sinus surgery
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygen Mask: Oxygen mask with oxygen flow 5 L/min will be given to allocated post general anesthesia patients. The incidence and causes of hypoxemia will be recorded.
  oxygen mask
- Oxygen Cannula: Oxygen cannula with oxygen flow 4 L/min will be given to allocated post general anesthesia patients. The incidence and causes of hypoxemia will be recorded.
  oxygen cannula
Period: Overall Study
Arm/Group | Oxygen Mask | Oxygen Cannula
Started | 250 | 250
Completed | 249 (One patient in oxygen mask received oxygen cannula) | 249 (1 patient in oxygen cannula group receive oxygen mask)
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients aged between 18-70 years who were scheduled for elective surgery under general anesthesia and had American Society of Anesthesiologists (ASA) physical status 1-3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxygen Mask | Oxygen Cannula | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.0) | 48.7 (13.8) | 48.65 (13.9)
Gender [Count of Participants; unit: Participants]
  Female | 180 | 161 | 341
  Male | 70 | 89 | 159
Region of Enrollment [Number; unit: participants]
  Thailand | 250 | 250 | 500

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hypoxemia in Both Groups
Description: Hypoxemia is defined as oxygen saturation < 94%. We record number of participants with hypoxemia in both groups
Time Frame: In PACU (1 hr after anesthesia)
Measure: Number; unit: number of participants
Arm/Group | Oxygen Mask | Oxygen Cannula
Number analyzed (Participants) | 250 | 250
number of participants | 0 | 0

2. Secondary Outcome: The Causes of Hypoxemia
Description: Causes of hypoxemia in each participant in PACU will be recorded
Time Frame: In PACU (1 hr after anesthesia)
Measure: Number; unit: causes of hypoxemia
Arm/Group | Oxygen Mask | Oxygen Cannula
Number analyzed (Participants) | 250 | 250
causes of hypoxemia | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 hour after anesthesia (in post-anesthesia care unit)
Description: Adverse events such as hypoxemia, re-intubation, unplanned ICU admission will be recorded. There were no serious adverse events.
Arm/Group | Oxygen Mask | Oxygen Cannula
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes